CLINICAL TRIAL: NCT01260415
Title: A Phase II Study of Perioperative Chemotherapy Plus Panitumumab in Patients With Colorectal Cancer Liver Metastases
Brief Title: A Study of Perioperative Chemotherapy Plus Panitumumab in Patients With Colorectal Cancer Liver Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMH DDP - CRCLM1
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: colorectal cancer; liver metastases; panitumumab; FOLFOX; Colorectal cancer with liver metastases
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Folfox/Folfiri, Panitumumab (Experimental): Eligible patients will recieved chemotherapy/panitumumab for 2 months (4 cycles) pre-operatively and 4 months post-operatively, plus a further 6 months of pantimumab post-chemotherapy
  Interventions: Drug: Panitumumab, Oxaliplatin, 5-FU

INTERVENTIONS:
Drug: Panitumumab, Oxaliplatin, 5-FU — * Panitumumab 6 mg / kg, given over 60 minutes
  * Oxaliplatin 85 mg / m2 combined with leucovorin 400 mg / m2, given over 2 hours OR
  * Irinotecan 180 mg / m2 , given over 90 minutes, concurrent with leucovorin 400 mg / m2, given over 90 minutes
  * 5FU 400 mg / m2, by bolus infusion
  * 5FU 2400 mg / m2, given over 46 hours

SUMMARY:
This is a phase II study to assess whether treatment with chemotherapy drugs FOLFOX (5-Fluorouracil (5FU), Oxaliplatin (Eloxatin) and Leucovorin (Folinic Acid)) or FOLFIRI (5-Fluorouracil (5FU), Irinotecan (Camptosar) and Leucovorin (Folinic Acid))and panitumumab before and after surgery can improve outcome in patients with liver metastases (the cancer has spread to other parts of the body such as the liver) that are resectable (can be surgically removed), from colorectal cancer that have a non mutant (wild-type) K-ras gene.

FOLFOX/FOLFIRI is an intravenous (given by vein) chemotherapy combination that is approved for colorectal cancer while panitumumab is also an intravenous drug and have been approved for treatment of refractory (not responding treatment) metastatic colorectal cancer whose cancers have the K-ras gene. These drugs are not approved for the treatment of colorectal cancer liver metastases (CRCLM) who can have surgery.

Patients will receive FOLFOX/FOLFIRI and panitumumab for four 2-week cycles before surgery. Surgery will be done no sooner than 4 weeks and no later than 8 weeks, after completion of the fourth cycle of chemotherapy.

If the liver metastases after the chemotherapy and surgery decreases or stops growing, then chemotherapy will be given after surgery. Treatments will start no sooner than 4 weeks, and no later than 12 weeks, after surgery. Patients will receive a maximum of 8 cycles of treatment with the combination of drugs and then receive panitumumab alone for a maximum of 12 cycles.

On treatment visits, patients will also have tests and procedures done. As part of the study, patients will provide archival tumor tissue and sample of tissue removed from surgery for K-ras testing. Patients will also be given the option of allowing the collected tissue for research (biomarker) studies and banking for future studies.

DETAILED DESCRIPTION:
Emerging data suggests that KRAS mutation is a strong predictor for resistance to EGFR antagonist therapy. In the KRAS wild-type cohort, the addition of EGFR antagonists to chemotherapy has been shown to improve RR and PFS. Improved response rate to neoadjuvant chemotherapy would be expected to improve surgical outcomes for patients with CRCLM. We therefore wish to test the hypothesis that the combination of FOLFOX/FOLFIRI and panitumumab, given perioperatively to patients with wild-type KRAS CRCLM will improve outcome, compared to historical control, in optimally resectable patients. As this patient population remains at high risk for recurrence post-chemotherapy, we also wish to explore the tolerability and efficacy of continued panitumumab monotherapy for an additional 6 months.

As opposed to most clinical trials for advanced colorectal cancer where the majority are treated with palliative intent, patients in this trial will all be treated aggressively with curative intent at the outset. There is also the additional benefit of assessment of tumor tissue after treatment with a biologic agent.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed colorectal cancer with available tissue to test for K-RAS mutation. Biopsy is required if no archived tissue is available. K-RAS mutation status must be confirmed prior to registration. Only patients with K-RAS wild-type cancers are eligible.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
* Patients must have resectable hepatic colorectal metastases.
* Patients may have synchronous unresected primary disease upon registration. Primary must be resectable, either at same laparotomy or at separate laparotomy from liver resection.
* Age >18 years.
* Patients must have Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
* Patients must have normal organ and marrow function as defined below:

leukocytes > 3,000/mcL absolute neutrophil count >1,500/mcL platelets >100,000/mcL hemoglobin > 90 g/L total bilirubin < 2 x upper limit of normal (< 1.5 x ULN for FOLFIRI), AST(SGOT) and ALT(SGPT)< 5 x upper limit of normal (< 3 x ULN for FOLFIRI);creatinine within normal institutional limits OR- creatinine clearance >50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal

* Appropriate imaging investigations, including CT or MRI of chest/abdomen/pelvis. Other scans if clinically indicated may be performed. All imaging studies must be performed within 28 days of study entry.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study and for a period of six months after cessation of study therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Patients must have had no previous systemic treatment in the adjuvant or metastatic setting within 6 months of registration.
* Patients may not have had prior treatment with an EGFR antagonist.
* Patients may not have a history of other malignancies, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid malignancies curatively treated with no evidence of disease for ≥ 5 years.
* Patients may not have extrahepatic metastatic disease. Patients who have had prior surgical resection for hepatic metastases or extrahepatic disease (eg. pulmonary metastases) are also excluded from this study.
* Patients may not have pre-existing chronic hepatic disease (eg. cirrhosis, chronic active hepatitis B or C)
* History of allergic reactions, or intolerance, attributed to compounds of similar chemical or biologic composition to 5-fluorouracil, oxaliplatin, or panitumumab.
* Patients being considered for irinotecan must not have a history of Gilbert's syndrome.
* Patients may not have uncontrolled inter-current illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with the agents used in this study. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Patients with active cardiovascular disease, i.e., unstable angina, New York Heart Association grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medications, or grade II or greater peripheral vascular disease. In addition, patients with arterial or venous thrombosis, myocardial infarction, and cerebral vascular accidents (stroke / transient ischemic attach (TIA)) within 6 months prior to study entry will be excluded.
* Patients with a history of interstitial pneumonitis or pulmonary fibrosis will be excluded.
* Organ allografts requiring immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To determine the 2 year disease-free survival rate in patients with resectable colorectal liver metastases treated with FOLFOX/FOLFIRI + panitumumab for 2 months pre-operatively and 4 months post-operatively, followed by panitumumab alone for 6 months. | 2-years post-therapy

SECONDARY OUTCOMES:
To evaluate the objective response rate (ORR) to preoperative FOLFOX/FOLFIRI plus panitumumab (by RECIST criteria) in patients with wild type KRAS. | until relapse
To evaluate the pathologic complete response rate. | until relapse
To determine overall survival and toxicity. | until death
To explore correlative biomarkers of clinical response (EGFR, PTEN, MET, BRAF and PI3KCA). | pre/post surgery
To explore for correlation between available tissue from biopsy, primary tumor and metastatic lesion with regards to aforementioned pathologic biomarkers. | pre/post surgery
To determine the incidence of hepatocellular damage (fibrosis, steatosis) in normal liver tissue induced by preoperative chemotherapy. | pre-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Welch, MD, Study Chair — London Regional Cancer Center; Sean Cleary, MD, Principal Investigator — Toronto General Hospital
Locations (4):
- Canada (4):
  - London Regional Cancer Centre, London, Ontario
  - The Ottawa Hospital Cancer Center, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario